CLINICAL TRIAL: NCT03543553
Title: From Brain Currents to Interpersonal Flow: Investigating the Social Processing Stream of Schizophrenia
Acronym: ecoval
Status: Not yet recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anja Vaskinn, Principal investigator, Oslo University Hospital
Other Study IDs: ecoval
Record Dates: First submitted 2018-04-17; First posted 2018-06-01 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Cognitive Impairment; Social Competence
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Social Skills

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SZ: Individuals with a diagnosis of schizophrenia
  Interventions: Other: This is not an intervention study
- HC: Healthy control participants
  Interventions: Other: This is not an intervention study

INTERVENTIONS:
Other: This is not an intervention study — This is not an intervention study

SUMMARY:
The overall objective of this project is to identify the neural signature of the impaired ability to relate socially seen in individuals with schizophrenia. A hypothesized path from the neural processes of social cognition, to social cognition assessed behaviorally, to real-life social interactions is examined. Secondary aims are to compare electrophysiological measures of high vs low level social cognition; to develop assessment methods of real-life behavior; and to increase the ecological validity of schizophrenia research. Much research within the field is devoid of personal meaning and interpersonal context. This project's use of personalized assessment allows for an ecologically valid approach to the social deficits of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia
* schizoaffective disorder

Exclusion Criteria

* diabetes
* Hyperthyroidism
* severe head trauma
* neurological disease

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with a diagnosis of schizophrenia will be compared to healthy control participants
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Neurophysiology: EEG | 1 day (when assessed)
  EEG mu suppression paradigm using point-light displays
Neurophysiology: ERP | 1 day (when assessed)
  ERP mentalizing paradigm (perspective taking)
Cognition | 1 day (when assessed)
  Matrics Consensus Cognitive Battery
Negative symptoms: clinician-rated | 1 day (when assessed)
  Positive and Negative Syndrome Scale (PANSS) 2. Objectively assessed using computerized software (FaceReader, PRAAT) of video-taped personal narratives produced by the participants
Negative symptoms: objective 1 | 1 day (when assessed)
  FaceReader
Negative symptoms: objective 2 | 1 day (when assessed)
  PRAAT
Social cognition: complex ToM | 1 day (when assessed)
  Movie for the Assessment of Social Cognition
Social cognition: low level ToM | 1 day (when assessed)
  The Hinting Task
Social cognition: facial emotion perception | 1 day (when assessed)
  Pictures of Facial Affect
Social cognition: body language reading | 1 day (when assessed)
  Emotion in Biological Motion test
Functioning | 1 day (when assessed)
  Social Functioning Scale (SFS). Seven scales that can be combined into a total score. Mean score in a schizophrenia population = 100, SD = 15. For both the seven scales and the total score.
Real-world behaviour | 1 day (when assessed)
  Day Reconstruction Method
Real-world social interactions | 1 day (when assessed)
  Video-ethnography

IPD SHARING:
Plan to Share IPD: No